CLINICAL TRIAL: NCT02679911
Title: Subject Adherence and Satisfaction for Treatment of Onychomycosis With Loceryl Nail Lacquer 5% Versus Ciclopirox Nail Lacquer
Brief Title: Treatment of Onychomycosis With Loceryl (Amorolfine) Nail Lacquer 5% Versus Ciclopirox Nail Lacquer
Acronym: LOOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR105082; 2015-001237-24 (EudraCT Number)
Record Dates: First submitted 2015-11-20; First posted 2016-02-11 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2018-02

CONDITIONS: Foot Dermatoses
Keywords: Onychomycosis
MeSH Terms: conditions — Foot Dermatoses; Onychomycosis

STUDY DESIGN:
Intervention Model Description: Intra-individual study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loceryl NL (Experimental): Amorolfine hydrochloride NL 5% to be applied once weekly for 12 weeks on all affected toenails of one foot
  Interventions: Drug: Loceryl NL
- Ciclopirox NL (Active Comparator): Ciclopirox NL 8% to be applied once daily for 12 weeks on all affected toenails of the opposite foot
  Interventions: Drug: Ciclopirox NL

INTERVENTIONS:
Drug: Loceryl NL — Topical over the entire toenail plate of all affected toenails, once weekly in the evening (at bed time) after filing down the affected toenails.
  Other Names: Loceryl Nail Lacquer
  Arms: Loceryl NL
Drug: Ciclopirox NL — Topical over the entire toenail plate of all affected toenails and surrounding skin, once daily in the evening (at bed time) after removing the free toenail edge and diseased toenails if needed
  Other Names: Ciclopirox Nail Lacquer
  Arms: Ciclopirox NL

SUMMARY:
The main objective of this study is to compare subject's compliance and satisfaction for two modes of treatment of toenails infection (Onychomycosis) with Loceryl Nail Lacquer (Loceryl NL) and Ciclopirox Nail Lacquer (Ciclopirox NL).

DETAILED DESCRIPTION:
A total of 20 subjects are to be included in 1 site in Germany.

Methodology:

Subjects will receive the following treatments on the right or left toenails:

* Loceryl Nail Lacquer to be applied once weekly for 12 weeks on all affected toenails of one foot.
* Ciclopirox Nail Lacquer to be applied once daily for 12 weeks on all affected toenails of the opposite foot.

ELIGIBILITY:
Inclusion Criteria:

* Subject with clinically Distal and Lateral Subungual Onychomycosis (DLSO) due to dermatophytes and/or yeast (including Candida) on at least one toenail of each foot at screening visit,
* Subject with less than 80% of the nail surface area with disease involvement and without matrix involvement, no dermatophytoma, streaks (spikes) or subungual hyperkeratosis > 2mm,
* Subjects with positive mycological results (direct microscopy and culture) for dermatophytes and/or yeasts (including Candida) at baseline,
* Subjects with same number of affected toenails on both feet or no more than one additional affected toenail on one of the feet,

Exclusion Criteria:

* Subject with a surgical, medical condition or clinically important abnormal physical findings, which, in the judgement of the investigator, might interfere with interpretation of the objectives of the study (i.e. lack of autonomy),
* Subjects with post-traumatic nail, lichen planus, eczema, psoriasis, or other abnormalities of the nail unit, which could affect/influence the subject's compliance of the investigational products, or mask the effects of treatment (cure),
* Subjects with known immunodeficiency, radiation therapy, immune suppressive drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Schaller, Principal Investigator — Universitäts-Hautklinik
Locations (1):
- Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects at screening had a mycological sampling of affected great toenail and for inclusion subjects shoud have both direct microscopy and culture results positive at Baseline
Groups:
- Loceryl NL and Ciclopirox NL: Loceryl Nail Lacquer to be applied once weekly for 12 weeks over the entire toenail plate of all affected toenails in the evening (at bed time) after filing down the affected toenails.
  Ciclopirox NL to be applied once daily for 12 weeks over the entire toenail plate of all affected toenails and surrounding skin in the evening (at bed time) after removing the free toenail edge and diseased toenails if needed
Period: Overall Study
Arm/Group | Loceryl NL and Ciclopirox NL
Started (This is an intraindividual study so only 20 subjecst are included in total) | 20 (Intra-individual study)
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Loceryl NL + Ciclopirox NL: Loceryl Nail Lacquer to be applied once weekly for 12 weeks over the entire toenail plate of all affected toenails in the evening (at bed time) after filing down the affected toenails.
  Ciclopirox NL to be applied once daily for 12 weeks over the entire toenail plate of all affected toenails and surrounding skin in the evening (at bed time) after removing the free toenail edge and diseased toenails if needed
Arm/Group | Loceryl NL + Ciclopirox NL
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  Germany | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent of "in Label" Adherent Subjects
Description: Percent of subjects having applied both treatments as instructed per labeling (once a week for Loceryl NL and once a day for Ciclopirox after 2 weeks)
Time Frame: Week 12
Population: Intention To Treat popoulation (ITT)
Measure: Number; unit: percentage of participants
Groups:
- Loceryl NL: Loceryl Nail Lacquer to be applied once weekly for 12 weeks over the entire toenail plate of all affected toenails in the evening (at bed time) after filing down the affected toenails.
- Ciclopirox NL: Ciclopirox NL to be applied once daily for 12 weeks over the entire toenail plate of all affected toenails and surrounding skin in the evening (at bed time) after removing the free toenail edge and diseased toenails if needed
Arm/Group | Loceryl NL | Ciclopirox NL
Number analyzed (Participants) | 20 | 20
percentage of participants | 85 | 60

2. Secondary Outcome: Percent of Subjects Satisfied to Very Satisfied With Each Study Treatment at Week 12
Description: Percent of subjects satisfied to very satisfied with both treatments (Loceryl nail lacquer and/or Ciclopirox nail lacquer) at week 12
Time Frame: Week 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Loceryl NL | Ciclopirox NL
Number analyzed (Participants) | 20 | 20
percentage of participants | 60 | 60

ADVERSE EVENTS:
Time Frame: During the study (12 weeks)
Groups:
- Loceryl NL + Ciclopirox NL: Loceryl Nail Lacquer to be applied once weekly for 12 weeks over the entire toenail plate of all affected toenails in the evening (at bed time) after filing down the affected toenails.
  Ciclopirox NL to be applied once daily for 12 weeks over the entire toenail plate of all affected toenails and surrounding skin in the evening (at bed time) after removing the free toenail edge and diseased toenails if needed
  Note: Adverse Events are not available for each intervention.
Arm/Group | Loceryl NL + Ciclopirox NL
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loceryl NL + Ciclopirox NL (N=20)
Nausea (Gastrointestinal disorders) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes